CLINICAL TRIAL: NCT01879436
Title: The Effect of Human Placental Explants and Pregnant Women Sera on Cancer Cells
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0053-13-MMC
Record Dates: First submitted 2013-06-10; First posted 2013-06-17 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Cancer
Keywords: Pregnancy, Placenta, Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Placentae will be collected and used in cell culture experiments for a week. Their proteins and RNA will be analyzed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pregnant women: Women during first trimester of pregnancy (age: 18-45)
  Group contain 50 healthy pregnant women, age 18-45. Sera will be taken from: 1. the same branula that will be introduced into the pregnant women as a routine during pregnancy termination procedure.2. from the vein of volunteered pregnant women which do not terminate pregnancy. First trimester placenta will be collected after pregnancy termination.
  The measure of outcome is composite and includes several changes:
  Changes in:
  * cell death (% from tested cells)
  * cell cycle (% cells in G1, G2 and S phases)
  * cell migration (% closure in Scratch test)
  * cell invasion (% cells passing through membrane in Transwell assay)
  * RNA repertoire (Fold change)
  * miRNA repertoire (Fold change) Investigators will not treat the women with any drug.
- Non pregnant women: Group contain 50 healthy women, age 18-45. Sera will be taken from the vein of the volunteered women. Investigators will not treat the women with any drug.

SUMMARY:
Maternal malignancy during pregnancy is estimated to occur in 1 out of 1000 pregnancies. Controversy exists regarding the effect of pregnancy on cancer prognosis. Gestational hormones and pregnancy-related growth factors may induce a more aggressive behavior in malignant cells. However, metastasis to the products of conception is rare. In the current study investigators wish to analyze the effect of placental explants on cancer cells (cervical, ovarian, thyroid, melanoma, lymphoma, leukemia and breast)phenotype (cell death, proliferation, migration , invasion), signaling pathway, mRNA, miRNA and protein expression.

DETAILED DESCRIPTION:
In the Oncogenetic laboratory cancer cells will be exposed to first trimester human placental explants or to serum collected from pregnant women. As a control cancer cells will be cultured alone or in the presence of sera collected from young (18-45) non pregnant women.

Placentae, 6-9 weeks gestational age, will be retrieved from terminated normal pregnancies. The placenta will be taken after pregnancy termination, thus, no harm will be caused for the women.

The sera will be collected from the women by an authorized physician. It will be taken from: 1. the vein of the non pregnant women and volunteered pregnant women. 2. from the same branula that will be introduced into the pregnant women as a routine during pregnancy termination procedure.

Following culture investigators will analyze the cancer cells phenotype (cell death, proliferation, migration, and invasion), signaling pathway, mRNA, miRNA and protein expression.

Sera will be collected from 50 pregnant women and 50 non pregnant women. Placentae will be collected from 50 pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Age 18-45.
* Pregnant (6-9 weeks) and non pregnant women.

Exclusion Criteria:

• Placentae that were destroyed during pregnancy termination.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women Age 18-45. Pregnant (6-9 weeks) and non pregnant women.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Cancer cell phenotype (in the laboratory) | Baseline, 24 hours and 72 hours
  The measure of outcome is composite and includes several changes:
  Changes in:
  * cell death (% from tested cells)
  * cell cycle (% cells in G1, G2 and S phases)
  * cell migration (% closure in Scratch test)
  * cell invasion (% cells passing through membrane in Transwell assay)
  * RNA repertoire (Fold change)
  * miRNA repertoire (Fold change)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lishner, MD, Principal Investigator — Meor Medical Center, Kfar-Saba, Israel
Locations (1):
- Oncogenetic Laboratory, Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Tartakover-Matalon S, Mizrahi A, Epstein G, Shneifi A, Drucker L, Pomeranz M, Fishman A, Radnay J, Lishner M. Breast cancer characteristics are modified by first trimester human placenta: in vitro co-culture study. Hum Reprod. 2010 Oct;25(10):2441-54. doi: 10.1093/humrep/deq227. Epub 2010 Aug 18. PMID 20719812